CLINICAL TRIAL: NCT03061799
Title: Efficacy and Safety of HPC-03(Extracts of Angelica Gigas Nakai, Cnidium Rhizome, and Cinnamon Bark) for Postmenopausal Symptom
Brief Title: Efficacy and Safety of HPC-03 for Postmenopausal Symptom
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jae Hoon Lee (Other)
Collaborators: Gachon University Gil Medical Center (Other); Daejeon University (Other)
Responsible Party: Sponsor-Investigator, Jae Hoon Lee, Cinical Fellow, Severance Hospital
Organization: Severance Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4-2016-0680
Record Dates: First submitted 2017-01-22; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Postmenopausal Period

STUDY DESIGN:
Intervention Model Description: This clinical trial will be conducted in parallel with the test group or the control group randomly assigned.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The product manufactured as clinical food and placebo are identical in shape, color and weight. In addition, clinical trial food should be labeled by affixing the same label with placebo so that it remains blind to both subjects and the investigator. Lot number of the label, includes reference number of the test food and reference number of the placebo together.
  Dispensing of food and placebo for clinical trials is handled by the management pharmacist.
  Clinical tester supplies clinical trial food corresponding the random assignment code assigned to subjects. Except inevitable cases such as occurrence of adverse events resulted by clinical food, the code will not be released until the end of the clinical trial. In case of deficiency or breakage of food for clinical trial, extra clinical food with unique code will provided to subjects, therefore maintain blinding.

ARMS (2):
- HPC-03 (Experimental): To experimental arm randomly assigned, HPC-03 will administrated twice a day , two capsules each time (total dose of HPC-03: 2g/day) for 12 weeks (84days).
  *(HPC-03: extracts of angelica gigas nakai, cnidium rhizome, and cinnamon bark.)
  Interventions: Dietary Supplement: HPC-03
- Placebo (Placebo Comparator): To control arm randomly assigned, placebo will administrated twice a day , two capsules each time for 12 weeks (84days).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: HPC-03 — HPC-03 is extracts of danggui (angelica gigas nakai), taeunggung (cnidium rhizome), and broilers (cinnamon bark).
  Other Names: angelica gigas nakai, cnidium rhizome, and cinnamon bark
  Arms: HPC-03
Dietary Supplement: Placebo — Placebo is constituted of crystalline cellulose(50.5%), corn starch(33.10%), caramel color(1.90%), anhydrous citric acid(1.25%), silicon dioxide(1.90%), carboxymethylcellulose calcium(6.25%), magnesium stearate(2.50%), and coater (3.10%).
  Arms: Placebo

SUMMARY:
In women, as the age increases, ovarian function is lost, resulting in the deficiency of female hormones, resulting in menopause, in which menstruation is permanently lost. The average age of menopause in Korean women is 49.7 years old, which is equivalent to 22.3% of the total female population. In addition, the increase in the number of women who experience early menopause due to environmental factors such as stress as a result of the increase in the number of women entering the society is also a major cause of the expansion of the market for menopausal women's health functional foods. Women's menopausal symptoms have been regarded as a natural process for everyone, but with the recent interest in health and the results of related studies, the perception that menopausal symptom management is necessary has spread.

In traditional medicine of far east asia, danggui (Angelica gigas Nakai), taeunggung (Cnidium Rhizome), and broilers (Cinnamon bark) have been commonly used for postmenopausal symptoms improvement. However, scientific evidence for these foods are lacking. Therefore, in this study the investigators tried to examine the efficacy and safety of extracts of angelica gigas nakai, cnidium rhizome, and cinnamon bark in postmenopausal symptoms. This study is designed as double-blinded placebo control study.

DETAILED DESCRIPTION:
The results of preclinical efficacy evaluation of HPC-03 (Angelica gigas Nakai complex extract) obtained by mixing materials mentioned above showed that increase of serum estrogen level and increase of bone mineral density (BMD) of femur due to ALP(Alkaline phosphatase ) inhibition, bone related index (BALP,bone-specific alkaline phosphatase ; CTX- 1,C-terminal telopeptide-1 ; Osteocalcin).

Therefore, the investigators aimed to confirm the safety and efficacy of HPC-03 (a complex extract of Angelica gigas Nakai) which has been confirmed in preclinical studies, on the improvement of menopausal symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Women 40 to 60 years old who have passed one year or more since the last menstrual period
2. Women with a kupperman index score of 20 or higher
3. Women who have agreed to participate in this trial before the start of the clinical trial and who have written an informed consent

Exclusion Criteria:

1. Women with a body mass index (BMI) greater than 30 kg / m2
2. Women using hormone preparations such as female hormones or similar hormone preparations (plant extracts, etc.) within 3 months
3. Women with a history of endometrial hyperplasia, uterine cancer, endometrial cancer, breast or breast disease, sex hormone related cancer
4. A woman with a history of severe migraine within the past 1 year, diagnosed with thromboembolism, cerebrovascular disease, myocardial infarction, unstable angina, or coronary angioplasty
5. Women with severe mental illnesses such as depression and anxiety disorder, or those currently taking psychotropic drugs such as antidepressants
6. Women with irregular uterine bleeding after 1 year of menopause
7. Patients with uncontrolled hypertension (160 / 100mmHg or higher, after 10 minutes of clinical test subjects)
8. Patients with diabetes whose blood sugar is not controlled (fasting glucose 180 mg / dL or diabetes mellitus within 3 months)
9. Those with uncontrolled thyroid disease (those who are considered to be able to participate in this trial by the tester can participate)
10. drug or alcohol abuser
11. If ALT(Alanine transaminase ) or AST(Aspartate transaminase) exceeds 3 times the normal upper limit of the research institute
12. If creatinine exceeds twice the upper limit of the normal level of research institute
13. Mammography / PAP smear If a clinically significant abnormality (Breast imaging-reporting and data system: BI-RADS category 0 or 3 or more, PAP smear is not abnormal up to ASCUS:atypical cells of undetermined significance) is confirmed (BI-RADS Category 0, )
14. If you have participated in another clinical trial within one month of the start of this trial or plan to participate in another clinical trial during the trial period
15. If the tester judges that the test is inappropriate for this clinical trial
16. Women using thyroid hormone preparations, clonidine, anticoagulants or antithrombotic agents (Warfarin, Clopidogrel, etc.) within 3 months
17. Women who took medicines or health functional foods related to women's menopause within a month

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2017-05 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Modified Kupperman Index score at 6 weeks and 12 weeks | At baseline, 6weeks and 12 weeks after administration of HPC-03 or placebo

SECONDARY OUTCOMES:
endometrial thickness measured by transvaginal ultrasonography | At baseline and 12 weeks after administration of HPC-03
serum estradiol (E2) | At baseline and 12 weeks after administration of HPC-03 or placebo
serum FSH (Follicular stimulating hormone) | At baseline and 12 weeks after administration of HPC-03 or placebo
  Follicular stimulating hormone

OTHER OUTCOMES:
serum alkaline phosphatase | At screening and 6weeks and 12 weeks after administration of HPC-03 or placebo
serum osteocalcin | At baseline and 6weeks and 12 weeks after administration of HPC-03 or placebo
Urine N-terminal cross-linker telopeptidase | At baseline, 6weeks and 12 weeks after administration of HPC-03 or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Seok Kyo Seo, M.D., Ph.D., Study Director — Department of Obstetrics and Gynecology, Yonsei University College of Medicine
Locations (1):
- Severance hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim SY, Seo SK, Choi YM, Jeon YE, Lim KJ, Cho S, Choi YS, Lee BS. Effects of red ginseng supplementation on menopausal symptoms and cardiovascular risk factors in postmenopausal women: a double-blind randomized controlled trial. Menopause. 2012 Apr;19(4):461-6. doi: 10.1097/gme.0b013e3182325e4b. PMID 22027944